CLINICAL TRIAL: NCT03435042
Title: A Hypnosis-based Group Intervention to Improve Quality of Life in Children With Cancer and Their Parents.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Isabelle Bragard, Lecturer, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hypnose enfant cancer
Record Dates: First submitted 2018-02-07; First posted 2018-02-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Self Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with cancer + their siblings (Experimental)
  Interventions: Behavioral: Self care + Hypnosis group
- Parents of children with cancer (Experimental)
  Interventions: Behavioral: Self care + Hypnosis group

INTERVENTIONS:
Behavioral: Self care + Hypnosis group — Our groupal intervention is divided into 6 monthly 2-hour sessions in which some self-hypnosis exercises are proposed to participants. Self-care techniques are also discussed (knowing our own needs, self-respect, assertiveness, coping with ruminations...) and homework assignments are proposed to participants, in order to foster positive change.

SUMMARY:
Background: A lot of children with cancer suffer from emotional distress, fatigue and relational difficulties. Their parents are also impacted by the disease: their responsibilities increase and they can feel more distressed and tired. Different psychological interventions designed for ill children and their parents seem to be efficient to improve their social functioning, coping strategies and well-being. However, more research is needed in this field. Hypnosis is often used in paediatric oncology, mostly to decrease procedure-related pain and distress. It has been used efficiently to improve the well-being of adults with cancer. This paper describes a pilot study designed to assess the feasibility and interest of a group intervention combining self-care and hypnosis for children with cancer and their parents, and a quasi-experimental protocol aimed at assessing the efficacy of this group intervention to improve the quality of life of children and their parents.

Methods: Our pilot study showed that our intervention was feasible and positive for the participants. To test the efficacy of the intervention, two groups will be set up: one with children with cancer and their interested siblings, and one with their parents. Data will be collected for each group before and after the intervention by questionnaires and a semi-structured interview.

Discussion: There is a growing interest in hypnosis in oncology settings. The results of this study should improve knowledge about the efficacy of a group intervention combining self-care and hypnosis to improve quality of life of children with cancer and their family.

ELIGIBILITY:
Inclusion Criteria:

* Children and their siblings:

  * To be 8 to 18 year-old
  * To suffer from cancer (all localisations, stage and treatments accepted) or to have a sibling who suffer from cancer
  * To speak french
* Parents:

  * To have a child who suffer from cancer
  * To speak french

Exclusion Criteria:

* /

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in children's quality of life | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  Self-assessment of children's quality of life. Measured with the Pediatric Quality of Life Inventory-Cancer Module (PedsQL-3.0-Cancer) and the Pediatric Quality of Life Inventory-Core Module (PedsQL-4.0-Core). Children with cancer answer to both questionnaires but their siblings only answer the PedsQL-4.0-Core.
Change in parents' conception of their child's quality of life | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  Parents' hetero-evaluation of the child's quality of life. Measured with the Parental version of the Pediatric Quality of Life Inventory-Cancer Module (PedsQL-3.0-Cancer) and the Parental version of the Pediatric Quality of Life Inventory-Core Module (PedsQL-4.0-Core).
Change in children's cancer-related fatigue | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  A sense of tiredness or exhaustion linked with cancer and its treatments, that is not alleviated by sleep. Measured with the Pediatric Functional Assessment of Chronic Illness Therapy-Fatigue (pedsFACIT-F) among children with cancer and their siblings .
Change in parents' fatigue | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  Measured with the Multidimensional Fatigue Inventory (MFI-20).

SECONDARY OUTCOMES:
Change in the family impact of the cancer | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  Impact of the child's health on the parents' quality of life and on the familily fonctioning. Measured with the Pediatric Quality of Life Inventory-Family Impact Module (PedsQL-2.0-Family Impact Module)
Change in parents' emotional distress | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  Anxiety and depression of the parents measured with the Hospital Anxiety and Depression Scale (HADS)
Change in parents' coping strategies | T0 (before the intervention), T1 (right after the intervention : 6 months later)
  The way parents cope adverses events. Measured with Ways of Coping Checklist (WWC-R)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elisabeth Faymonville, Study Director — Centre Hospitalier Universitaire de Liege
Locations (1):
- University Hospital of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregoire C, Chantrain C, Faymonville ME, Marini J, Bragard I. A HYPNOSIS-BASED GROUP INTERVENTION TO IMPROVE QUALITY OF LIFE IN CHILDREN WITH CANCER AND THEIR PARENTS. Int J Clin Exp Hypn. 2019 Apr-Jun;67(2):117-135. doi: 10.1080/00207144.2019.1580965. PMID 30939086